CLINICAL TRIAL: NCT03852823
Title: An Open, Multi-dose, Dose Escalation and Cohort Expansion, Phase Ⅰ Study of the Recombinant Human Anti-PD-1 Monoclonal Antibody in Patients With Advanced Tumours.
Brief Title: Study of Recombinant Human Anti-PD-1 Monoclonal Antibody in Patients With Advanced Tumours
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SG001201801
Record Dates: First submitted 2019-02-20; First posted 2019-02-25 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Advanced Solid Tumours; Cervical Cancer; Malignant Mesothelioma; Lymphoma; Non-Small-Cell Lung Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Mesothelioma, Malignant; Lymphoma; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SG001 (Experimental): Recombinant Human Anti-PD-1 Monoclonal Antibody
  Interventions: Drug: SG001

INTERVENTIONS:
Drug: SG001 — Phase Ia: Subjects will receive intravenous infusion of SG001 following a sequential dose escalation design (1mg/kg, 3mg/kg and 10mg/kg). Dose limited toxicity (DLT) will be observed within 21 days after the first administration, then subjects can continuously receive SG001 every 2 weeks until confirmed progression, unacceptable toxicity, or withdrawal from the trial. Phase Ib: Subjects will receive intravenous infusion of SG001 at the dose of 240 mg every 2 weeks until confirmed progression, unacceptable toxicity, or withdrawal from the trial.
  Other Names: Recombinant Human Anti-PD-1 Monoclonal Antibody

SUMMARY:
This study is an open, multi-dose, dose escalation and cohort expansion, phase Ⅰ study to investigate the safety, tolerability, efficiency, pharmacokinetics, immunogenicity of SG001 in subjects with advanced tumours.

DETAILED DESCRIPTION:
Phase Ⅰa: open, multi-dose, dose escalation. Phase Ⅰb: open, fixed-dose, cohort expansion.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 on the day of signing informed consent.
* Phase Ⅰa: Histologically/cytologically confirmed diagnosis of advanced solid tumor, and failure of standard anti-tumor treatment (disease progression or intolerance), or no standard treatment or rejection of standard treatment.

Phase Ⅰb:

Cohort A: Histologically or cytologically documented locally-advanced, relapsed or metastatic solid malignancy with PD-L1 positive and/or deficiency in mismatch repair (dMMR) / Microsatellites instability-High (MSI-H) and/or EBV positive, and has failed at least first line standard therapy or for which standard therapy is not tolerated.

Cohort B: Histologically documented relapsed or metastatic uterine cervical cancer and has failed at least first line standard therapy or for which standard therapy is not tolerated.

Cohort C: Histologically documented malignant mesothelioma, and has failed to pemetrexed-based chemotherapy or chemotherapy is not tolerated.

Cohort D: Histologically documented relapsed or refractory lymphoma, and has failed at least 2 lines standard therapy, including radiotherapy or autologous hematopoietic stem cell transplantation.

Cohort E: Histologically or cytologically documented non-small cell lung cancer without EGFR or ALK gene mutation, and has failed at least first line standard therapy or for which standard therapy is not tolerated.

* Solid tumor except malignant pleural mesothelioma will be assessed by RECIST 1.1, malignant pleural mesothelioma will be evaluated by Modified RECIST for malignant pleural mesothelioma, and lymphoma will be assessed by Lugano criteria (2014). All the subjects should have at least one measurable lesion in CT or MRI test.
* If subjects have received anti-tumor therapies before, the toxicity severity must decrease to ≤ Grade1 evaluated by CTCAE 5.0, except for residual alopecia.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has a predicted survival period ≥ 3 months.
* Demonstrate adequate organ function as defined below(No anticoagulants or other drugs affecting clotting function were used within 14 days prior to the first administration. No blood transfusions were performed, no hematopoietic stimulators were used, and no drugs were used to correct blood cell counts). a) Hemoglobin (HGB)≥9 g/dL;b)Absolute neutrophil count (ANC) ≥1.5×109/L;c)Platelets ≥75×109/L;d) Serum total bilirubin (TBIL) ≤ 1.5 X upper limit of normal ULN (Subjects with Gilbert's syndrome can be up to 3 x ULN);e) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 X ULN or ≤5 X ULN for subjects with hepatocellular carcinoma and liver metastases;f)Serum creatinine ≤1.5 X ULN or Creatinine clearance (CCr) ≥ 50mL/min;g)International Normalized Ratio (INR) and activated partial thromboplastin time (APPT) ≤1.5 X ULN.
* From signing the informed consent form to 6 months after last dose of investigational drug, subjects of childbearing potential should be willing to use reliable contraceptive methods.

Exclusion Criteria:

* History of allergic reactions attributed to any monoclonal antibody, and uncontrolled history of allergic asthma.
* Subjects with primary central nervous system tumor, or symptomatic/untreated central nervous system metastases (except for residual signs or symptoms related to CNS treatment, those with stable or improved neurological symptoms at least 2 weeks before inclusion can be included)
* Patients with any autoimmune disease, i.e., but not limited to, subjects with well-controlled type I diabetes, well-controlled hypothyroidism with hormone replacement therapy, skin diseases (such as vitiligo, psoriasis, or hair loss) without systemic treatment, or who are not expected to relapse without external triggers.
* History of primary immunodeficiency
* Patients with serious cardiovascular diseases, such as grade 2 or above heart failure, previous myocardial infarction within 3 months, poorly controlled arrhythmias or unstable angina pectoris, as rated by New York Heart Association;.
* Has history of Interstitial Lung Disease or non-infectious pneumonitis. (Patients caused by radiotherapy are eligible).
* Prior therapy with an anti-PD-1, anti-PD-L1,or anti CTLA-4 antibody ( any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
* Immune-related adverse events of grade 3 or higher（CTCAE 5.0）after immune therapy.
* Have received allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
* Any active infection requiring systemic treatment by intravenous infusion within 14 days prior to screening.
* Have received major surgery or radical radiotherapy within 28 days, or palliative radiotherapy within 14 days, or radiological agents (strontium, samarium, etc.) within 56 days prior to screening.
* Have received systemic anti-tumour therapy 28 days before the first dose, including but not limited to chemotherapy, immunotherapy, macromolecular targeted therapy, and biological therapy (tumour vaccine, cytokines or growth factors controlling cancer); Patients who received small-molecule targeted and oral fluorouracil therapy within 14 days before the first dose (or 5 half-life, whichever is longer); Patients who received mitomycin C and urea nitrite within 6 weeks before the first dose.
* Live attenuated vaccine should be given within 14 days before screening or during the study period
* Have received Chinese herbal medicine or Chinese patent medicine with anti-tumor activity within14 days prior to the screening.
* Have received whole blood transfusion or blood component transfusion within 14 days prior to screening.
* Have a history of active tuberculosis or tuberculosis.
* Active hepatitis B virus infection or syphilis, or hepatitis C virus antibody or human immunodeficiency virus (HIV) antibody positive.
* Have participated other clinical trials and received related investigated drugs within 28 days prior to the first dose of study drug.
* Pregnant or lactating women; Or the blood pregnancy test of women at child-bearing age is positive during screening.
* Have received systemic corticosteroids (at doses equivalent to or greater than 10 mg/day of prednisone) or other immunosuppressive drugs within 14 days prior to the first dose of study drug.
* Other conditions that may increase the risk of drug use in the study, or interfere with the interpretation of the study results, or affect the compliance of the study, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2019-05-23 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of SG001 by assessing the percentage of participants who experience a dose-limiting toxicity (DLT) | Phase Ⅰa: 21 days
  To investigate the safety and tolerance profile tolerance profile of SG001 in subjects with advanced solid tumors
Objective response rate (ORR) in solid tumor（The ORR of cohort B, C, and E will be evaluated by Independent Review Committee）. | Phase Ⅰb: From date of first drug administration until the date of first documented progression of disease or the date of death or the date of lose to follow-up, which occurs first, assessed up to 2 years.
  To investigate the efficiency of SG001 in subjects with advanced solid tumors
Safety of SG001 in patients with advanced tumors. | Phase Ⅰb: From signing informed consent form (ICF) to 90 days after the last dose of study drug or initiation of a new therapy for cancer, which occurs first.
  To investigate the safety of SG001 in advanced tumors.

SECONDARY OUTCOMES:
The pharmacokinetic parameters of SG001, such as Cmax, AUC, t1/2 tmax, Vss, CL (clearance rate) etc. | Phase Ⅰa: At the end of cycle 7（every cycle is 14 days，except cycle 1 is 21 days）; Phase Ⅰb: At the end of cycle 13 （every cycle is 14 days）.
  The pharmacokinetics(PK) profile of SG001.
The ORR of cohort B, C, and E, which will be evaluated by investigators. | From date of first drug administration until the date of first documented progression of disease （PD） or the date of death or the date of lose to follow-up, which occurs first, assessed up to 2 years.
  The efficiency of SG001.
The ORR of cohort D, which will be evaluated by Lugano criteria 2014. | From date of first drug administration until the date of first documented progression of disease （PD） or the date of death or the date of lose to follow-up, which occurs first, assessed up to 2 years.
  The efficiency of SG001.
DOR (duration of response). | From the date of first documentation of confirmed CR（complete response）/PR（partial response） to the date of first documentation of PD or the date of death from any cause or the date of lose to follow-up, which occurs first, assessed up to 2 years.
  The efficiency of SG001.
DCR (disease control rate). | DCR is defined as the percentage of patients with best overall response of CR, PR, or SD（stable disease）, which will be assessed up to 2 years.
  The efficiency of SG001.
TTP (time to progression). | From the date of first drug administration to the date of first documentation of PD, assessed up to 2 years.
  The efficiency of SG001.
PFS (free-progression survival). | From date of first drug administration until the date of first documented progression of disease （PD） or the date of death, which occurs first, assessed up to 2 years.
  The efficiency of SG001.
OS (overall survival). | From date of first drug administration until the date of death, assessed up to 2 years.
  The efficiency of SG001.
Immunogenicity of SG001. | From the first dose of study drug to 28 days after its last dose.
  The immune profile of SG001.
The activated T cell receptor occupancy. | Phase Ⅰa: At the end of cycle 7（every cycle is 14 days，except cycle 1 is 21 days）; Phase Ⅰb: At the end of cycle 13 （every cycle is 14 days）.
  The pharmacodynamics of SG001.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, PhD, Principal Investigator — Shanghai East Hospital; Lingying Wu, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Caicun Zhou, PhD, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Fang J, Jiang O, Li W, Lin J, Fang M, Li Q, Zhao W, Wang K, Shi H, Chen Z, Yu J, Xing X, Zhao M, Liu A, Wang W, Han Z, Xiang S, Zhang X, Li J, Zhou C. Phase 1b Multicenter Study of SG001, a Humanized Anti-PD-1 Antibody, in Patients with Advanced Solid Tumors. Drug Des Devel Ther. 2025 Nov 24;19:10423-10435. doi: 10.2147/DDDT.S546663. eCollection 2025. PMID 41321671